CLINICAL TRIAL: NCT00179673
Title: A Phase II, Multicenter, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of Single-Agent Lenalidomide (Revlimid®, CC-5013) in Subjects With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Lenalidomide (Revlimid®, CC-5013) in Subjects With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Prologue Research International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NHL-001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: NHL; CC5013; Non-Hodgkins Lymphoma; revlimid; cc-5013; celgene
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental): Participants received single-agent lenalidomide 25 mg orally once daily on Days 1 to 21 of every 28-day cycle for up to 52 weeks or until disease progression developed.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid; CC-5013

SUMMARY:
Subjects who qualify will receive lenalidomide daily on days 1-21 of every 28-day cycle. Treatment will continue for up to 52 weeks or until disease progression; subjects who achieve a Complete Response (CR) will receive an additional 2 cycles of treatment prior to discontinuation. Subjects will be followed for progression free survival following discontinuation from the treatment phase

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age greater than or equal to 18 years at the time of signing the informed consent form
3. Able to adhere to the study visit schedule and other protocol requirements
4. Biopsy-proven non-Hodgkin's lymphoma
5. Indolent lymphoma the following histologies are acceptable: a. Follicular center lymphoma, grades 1, 2; b. Extranodal marginal zone B-cell lymphoma of Mucosa associated lymphoid tissue (MALT) type, c. Nodal marginal zone B-cell lymphoma d. Splenic marginal zone B-cell lymphoma, e. Small lymphocytic lymphoma (SLL), f. Lymphoplasmacytoid lymphoma
6. Relapsed or refractory to previous therapy for lymphoma. Participants must have received at least one prior treatment regimen such as radiation, immunotherapy, chemotherapy, or radioimmunotherapy, and be ineligible or unwilling to undergo an autologous stem cell transplant. There is no limit on the number of prior therapies
7. Participants must have measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
9. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.

Exclusion Criteria:

1. Any of the following laboratory abnormalities

   1. Absolute neutrophil count (ANC) <1,500 cells/mm^3 (1.5 x 10^9/L)
   2. Platelet count <100,000/mm^3 (100 x 10^9/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamic-pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) >5.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
2. Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. All participants with Central Nervous System (CNS) disease with the exception of those subjects whose CNS disease has been treated with chemotherapy, radiotherapy or surgery and remains asymptomatic, with no active CNS disease, as shown by lumbar puncture, computerized tomography (CT) scan or Magnetic resonance imaging (MRI), for at least 6 months.
4. Prior history of malignancies other than non-Hodgkin's lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the participant has been free of the disease for > or equal to 1 year.
5. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from signing the informed consent form.
6. Known positive for human immunodeficiency virus (HIV).
7. Pregnant or lactating females.
8. Prior > or equal to grade 3 allergic reaction/hypersensitivity to thalidomide.
9. Prior > or equal to grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
10. Prior use of lenalidomide.
11. Use of any standard or experimental anti-cancer drug therapy within 28 days of day 1 of study drug therapy.
12. Known active Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Alta Bates Cancer Center, Berkeley, California
  - Pacific Coast Hematology/Oncology Medical Group, Onc., Fountain Valley, California
  - Rush University Medical Center, Chicago, Illinois
  - Harvard University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - New York Medical Center, MBCCOP, The Bronx, New York
  - Signal Point Hematology/Oncology, Middletown, Ohio
  - Swedish Cancer Institute, Seattle, Washington
  - Gunderson Clinic, Ltd., La Crosse, Wisconsin
- Canada (4):
  - BC Community Oncology Trialist, Burnaby, British Columbia
  - BC Community Oncology, North Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: Participants received single-agent lenalidomide 25 mg orally once daily on Days 1 to 21 of every 28-day cycle for up to 52 weeks or until disease progression developed, lenalidomide treatment was discontinued for any reason, or the study was terminated.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 43
Received Study Drug | 43
Completed | 0 (Completed refers to participants ongoing in the study at the time of analysis.)
Not Completed | 43
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 15
Not completed — Withdrawal by Subject | 3
Not completed — Death | 4
Not completed — Other Observations and options | 14

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.95)
Age, Customized [Number; unit: participants]
  <65 years | 24
  65 - 75 | 10
  >75 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37
  Black | 4
  Hispanic | 0
  Asian/Pacific Islander | 1
  American Indian/Alaska Native | 0
  Other = Unspecified | 1
NHL Duration [Mean (Standard Deviation); unit: years] | 5.6 (4.38)
Non-Hodgkin's Lymphoma (NHL) Histology [Number; unit: participants] — I: The lymphoma is in only 1 lymph node area or 1 area of a single organ outside the lymph system. II: The lymphoma is in 2 or more groups of lymph nodes on the same side of the diaphragm, or extends from a single group of node(s) into a nearby organ. III: The lymphoma is found in lymph node areas on both sides of the diaphragm, or may also have spread into an area or organ next to the lymph nodes, the spleen, or both. IV: The lymphoma has spread outside the lymph system into an organ that is not next to an involved node or has spread to bone marrow, liver, brain, spinal cord or the pleura.
  participants
    Follicular lymphoma grade 1 or 2 | 22
    Small Lymphocytic lymphoma | 18
    Nodal marginal-zone B-cell lymphoma | 2
    Extranodal marginal-zone B-cell type (MALT) | 1
Non-Hodgkin's Lymphoma (NHL)-Stage [Number; unit: participants] — I: The lymphoma is in only 1 lymph node area or 1 area of a single organ outside the lymph system. II: The lymphoma is in 2 or more groups of lymph nodes on the same side of the diaphragm, or extends from a single group of node(s) into a nearby organ. III: The lymphoma is found in lymph node areas on both sides of the diaphragm, or may also have spread into an area or organ next to the lymph nodes, the spleen, or both. IV: The lymphoma has spread outside the lymph system into an organ that is not next to an involved node or has spread to bone marrow, liver, brain, spinal cord or the pleura.
  participants
    Stage I | 1
    Stage II | 11
    Stage III | 6
    Stage IV | 25
International Prognostic Index (IPI)] [Number; unit: participants] — A clinical tool to aid in predicting the prognosis of patients with NHL. One point is assigned for each of the following risk factors: • Age greater than 60 years • Stage III or IV disease • Elevated serum lactate dehydrogenase • ECOG performance status of 2, 3, or 4 • 1 extranodal site The sum of the points allotted correlates with the following risk groups: Low risk (0-1 points): 5-year survival of 73%; Low-intermediate risk (2 points): 5-year survival of 51%; High-intermediate risk (3 points): 5-year survival of 43%; High risk (4-5 points): 5-year survival of 26%.
  participants
    Low (0 to 1) | 14
    Low/Intermediate (2) | 15
    High/Intermediate (3) | 6
    High (4 to 5) | 8
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG-Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determines appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = fully active, no restrictions; | 27
    1 = restricted but ambulatory and capable of light | 12
    2 = ambulatory and capable of self care but unable | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Response was defined as participants with a complete response (CR), unconfirmed complete response (Cru) or partial response (PR), assessed using the International Workshop Lymphoma Response Criteria (IWLRC) and based on best responses as determined by the investigator. CR: Complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of any disease-related symptoms, and normalization of biochemical abnormalities. Cru: Criteria for CR above but with 1 or more of the following: • A residual lymph node mass > 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of diameters (SPD) • Indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia). PR: ≥ 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD.
Time Frame: From enrollment through study completion. Median duration on study was 4.4 months with a maximum of 32 months
Population: Intent-to-treat (ITT) population, which included all enrolled patients who received at least 1 dose of study drug. Patients who dropped out without having a response assessment or who had a response after they had received other anti-cancer treatments were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 43
percentage of participants | 23.3 [11.8 to 38.6]

2. Secondary Outcome: Percentage of Participants With Tumor Control
Description: Tumor control was defined as participants with a complete response, unconfirmed complete response, partial response or stable disease (SD), assessed using the International Workshop Lymphoma Response Criteria (IWLRC) and based on best responses as determined by the investigator. SD was defined as a response less than a PR (see above) but not Progressive Disease (PD). PD was defined as • ≥ 50 % increase from nadir in the SPD of any previously identified abnormal node for partial responders or non-responders. • Appearance of any new lesion during or at the end of therapy.
Time Frame: From enrollment through study completion. Median duration on study was 4.4 months with a maximum of 32 months
Population: Intent-to-treat (ITT) population. Patients who dropped out without having a response assessment or who had a response after they had received other anti-cancer treatments were considered non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 43
percentage of participants | 60.5 [44.4 to 75.0]

3. Secondary Outcome: The Duration of Response
Description: The duration of response was calculated as the first response assessment demonstrating evidence of at least a partial response to the first documentation of progressive disease (as determined by computed tomography scan) or death due to NHL, whichever occurred first. For participants without documentation of progression, the duration of response was censored at the last date of tumor assessment indicating no progression. Median was based on the Kaplan-Meier estimate.
Time Frame: From enrollment through study completion. Median duration on study was 4.4 months with a maximum of 32 months
Population: Includes participants with a response to treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 10
months | NA [15.5 to NA] — The median was not reached due to the low number of events.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from the start of study drug therapy to the first observation of disease progression or death due to any cause, whichever came first. Participants who withdrew for any reason or received another NHL therapy including stem cell transplantation without documented progressive disease were censored on the date of their last adequate response assessment indicating no progression (or last adequate assessment prior to receiving other NHL therapy). Participants who were still active without progressive disease at the time of the data cut-off date were censored on the date of their last adequate response assessment.
Time Frame: From enrollment through study completion. Median duration on study was 4.4 months with a maximum of 32 months
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 43
months | 4.4 [2.5 to 10.4]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The Investigator determined the relationship between the administration of study drug and the occurrence of an AE as suspected if the temporal relationship of the adverse event to study drug administration made a causal relationship possible, and other drugs, therapeutic interventions, or underlying conditions did not provide a sufficient explanation for the observed event. The Investigator graded the severity of AEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria and the following scale: • Grade 1 = Mild • Grade 2 = Moderate • Grade 3 = Severe • Grade 4 = Life threatening • Grade 5 = Death A Serious AE is defined as any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or constitutes an important medical event.
Time Frame: From the start of study drug through 30 days after the last dose of study drug. Maximum time on study drug was 13.8 months.
Population: Safety Population, which includes all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 43
participants
  At least one Adverse Event (AE) | 42
  ≥ 1 AE related to study drug | 37
  Grade (GR) 3-5 AE | 27
  Grade 3-5 AE related to study drug | 24
  Serious adverse event (SAE) | 18
  SAE related to study drug | 10
  AE leading to discontinuation of study drug | 9
  Related AE leading to study drug discontinuation | 5
  AE leading to dose reduction or interruption | 27

ADVERSE EVENTS:
Time Frame: From the start of study drug through 30 days after the last dose of study drug. Maximum time on study drug was 13.8 months
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 18/43
Other Adverse Events (participants affected / at risk) | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=43)
Anemia Not Otherwise Specified (NOS) (Blood and lymphatic system disorders) | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal Pain NOS (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea NOS (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Sepsis NOS (Infections and infestations) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Asthenia (General disorders) | 2 — General disorders and administration site conditions
Fatigue (General disorders) | 2 — General disorders and administration site conditions
Chest Discomfort (General disorders) | 1 — General disorders and administration site conditions
Oedema Peripheral (General disorders) | 1 — General disorders and administration site conditions
Leukocytosis (Blood and lymphatic system disorders) | 1
Gastrointestinal Obstruction NOS (Gastrointestinal disorders) | 1
Intestinal Fistula (Gastrointestinal disorders) | 1
Small Intestinal Obstruction NOS (Gastrointestinal disorders) | 1
Pneumonia NOS (Infections and infestations) | 2
Clostridial Infestion NOS (Infections and infestations) | 1
Infection NOS (Infections and infestations) | 1
Somnolence (Nervous system disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Airways Disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=43)
Fatigue (General disorders) | 20
Oedema Peripheral (General disorders) | 4
Pain NOS (General disorders) | 4
Pyrexia (General disorders) | 4
Constipation (Gastrointestinal disorders) | 13
Diarrhoea NOS (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 8
Abdominal Pain NOS (Gastrointestinal disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Leukopenia NOS (Blood and lymphatic system disorders) | 10
Anaemia NOS (Blood and lymphatic system disorders) | 7
Haemoglobin Decreased (Investigations) | 8
Neutrophil Count Decreased (Investigations) | 8
Alanine Aminotransferase Increased (Investigations) | 5
Blood Alkaline Phosphatase NOS Increased (Investigations) | 4
White Blood Cell Count Decreased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 3
Platelet Count Decreased (Investigations) | 3
Rash NOS (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 5
Night Sweats (Skin and subcutaneous tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 5
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 6
Tumour Flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.